CLINICAL TRIAL: NCT04036565
Title: The Sunlight Improves Depression in Stroke Patients
Brief Title: The Sunlight Exposure Therapy on the Improvement of Depression and Quality of Life in Post-stroke Patients
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-09-001CC
Record Dates: First submitted 2019-07-26; First posted 2019-07-29 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Depression
Keywords: Sunlight; depression; daily active function; stroke
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The experimental group: The first post-test measurements were taken right after the participants completed the sunlight therapy (two to four weeks after the start of the intervention), and the second post-test measurements were taken one month after the intervention was completed (six to eight weeks after the start of the intervention).
  Interventions: Behavioral: sunlight therapy
- The control group: Standard care.The first and second post-test measurements were taken two and six weeks, respectively, after they started receiving standard care.

INTERVENTIONS:
Behavioral: sunlight therapy — Exposed to sunlight for at least 30 minutes per day, at least 14 days of exposure duration of 4 weeks.
  Groups: The experimental group

SUMMARY:
Chronic diseases has been the leading causes of death in 2015 to 2017 based on the National database. In particular, cerebrovascular disease was the third in 2015, the fourth in 2016 and 2017. In the Statistical Office of the Ministry of Health and Welfare (2016, 2017,2018). Previous studies have suggested that nearly 30% of the stroke victims present with signs of depression within the first 5 years of illness. Since post-stroke depression significantly affects the patient both physically and psychologically, the emotional disturbances impede the progress and effectiveness of rehabilitation. Regarding the non-pharmacological treatment of melancholia, the phototherapy has been used to treat psychological, behavioral or emotional disorders with satisfactory outcomes.Furthermore, many studies has suggested that artificial light should mimic natural sunlight to reach optimal effect. The benefit of sunlight in human wellbeing has been well documented, therefore we intend to utilize sunlight therapy for stroke patients in order to improve their physical and mental health.

DETAILED DESCRIPTION:
This study is an experimental interventional study for two groups with pretest and posttest analysis. The subjects of the study met the inclusion criteria and were recruited by intention sampling method. They were randomly assigned to the experimental group and the control groups. This is a single-blind study with sunlight exposure as intervention. Appropriate clothing, skin protection measures were given. The calf portion of feet, forearms and hands were exposed to sunlight for at least 30 minutes per day, at least 14 days of exposure with intensity at least 10000lux over duration of 4 weeks. A total of 46 patients were recruited and 4 have lost follow up. 21 patients from each group have completed the study. The research tools include: depression status (Taiwanese depression scale,TDS), physical activity function (Barthel Index), the severity of cognitive function (mini-mental state examination,MMSE) and severity of stroke (National institutes of health stroke scale,NIHSS). Each patient was evaluated 3 times during the study: on the day of enrollment (pre-test), 2 to 4 weeks since enrollment (1st post-test) and 6-8 weeks after enrollment (2nd post-test). Statistical analysis was performed with the following variables: depression, cognitive function (MMSE), severity of stroke (NIHSS) and the Barthel Index for daily function.

The participants in the experimental and control groups were subjected to a pre-test measurement after they were recruited. For the experimental group, the first post-test measurements were taken right after the participants completed the sunlight therapy (two to four weeks after the start of the intervention), and the second post-test measurements were taken one month after the intervention was completed (six to eight weeks after the start of the intervention). For the control group, the first and second post-test measurements were taken two and six weeks, respectively, after they started receiving standard care.

At the start of intervention, the researchers conducting this study instructed the experimental group to fill out a sunshine exposure duration record sheet. The participants used symbols on the record sheet to indicate the day's weather, such as sunny, partly sunny, and cloudy and rainy. Sunshine records were excluded on cloudy and rainy days, while records were taken on partly sunny days with sufficient sunshine, and participants had to expose themselves outdoors to the sun in an outdoor environment; they were not allowed to expose themselves to the sun from an indoor environment through glass. Participants had to take appropriate protective measures on their own beforehand, such as wearing breathable clothing, visors or sunglasses, and applying sunblock. Throughout the implementation of the sunlight therapy, participants were allowed to rest and drink in shady areas if they had any discomforts (dizziness, hyperthermia), so as to avoid overexposure to sunlight. If they had a burning skin sensation or itchy skin, they were allowed to rinse their skin with cold water, iced water, or ice cubes, or to apply ice cubes on their skin for three to five minutes, so as to lower their skin temperature and alleviate skin allergies. They were advised to call for a medical examination or to contact the researchers if their symptoms persisted.

ELIGIBILITY:
Inclusion Criteria:

* Participants also had to meet at least two of the Diagnostic and Statistical Manual(DSM)-IV diagnosis criteria for minor depression, dejection, or dysthymia, and had to be conscious and capable of expressing themselves. Participants had to be aged 20 or above, able to converse in or be literate in Mandarin or Taiwanese, and agree, after being asked to provide consent, to participate in this study.

Exclusion Criteria:

* Patients with a NIHSS score higher than 16 (severe stroke); patients with stroke caused by cancer metastasis; stroke patients with cancer comorbidity; and patients who were on dialysis, pregnant, mentally-challenged, or suffering from severe cognitive disabilities.

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants had to be verified one-month post-stroke patients in stable condition, with an NIHSS score of not more than 15 (minor or moderate stroke).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
depression status (Taiwanese depression scale, TDS) | 8-12weeks
  change depression status. Assess the feeling of body and mood within 7 days. Those who are above 19 will be considered as those with severe depression. 15-18 is divided into depression points to the critical point. 9-14 is divided into emotional ups and downs.
physical activity function (Barthel Index) | 8-12weeks
  improved physical activity function. The total score of the scale is between 0 to 100 points. The higher the score, the better the activity Can be re-evaluated at different times, compare the difference in scores to determine whether daily life function is progressing or regressing

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 8-12weeks
  change stroke severity. The total score of the scale is between 0 to 38 points stroke severity was categorized as minor (NIHSS = 0 to 6), moderate (NIHSS = 7 to 15), and severe (NIHSS = 16 to 38)

OTHER OUTCOMES:
cognitive status (mini-mental state examination,MMSE). | 8-12weeks
  change cognitive status. A total of 11 evaluation projects. Can be divided into four parts including orientation, language, attention and memory.
  The content includes an assessment of the orientation, message acceptance, attention and arithmetic skills, short-term memory, language (reading, writing, naming, understanding, etc.) of the current time and place.
  The highest score is 30 points, 0-23 is abnormal, and 24 points is normal.

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Yen Chen, Study Director — School of Nursing, National Taipei University of Nursing and Health Sciences.
Locations (1):
- Su-Jen Wang, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Sunlight therapy intervention: The sun had to be bright and visible during the day, with an illuminance of 10,000 lux and above (Chang et al., 2011). Participants were required to employ appropriate protective measures when directly exposing their forearms or calves under the sun for an accumulated minimum of 30 minutes per day, for a total of 14 days in four weeks.

REFERENCES:
- [Result] West A, Jennum P, Simonsen SA, Sander B, Pavlova M, Iversen HK. Impact of naturalistic lighting on hospitalized stroke patients in a rehabilitation unit: Design and measurement. Chronobiol Int. 2017;34(6):687-697. doi: 10.1080/07420528.2017.1314300. Epub 2017 Apr 21. PMID 28430522